CLINICAL TRIAL: NCT02793453
Title: Antimicrobial Peptides in Periodontitis : a Pilot Study
Brief Title: Antimicrobial Peptides in Periodontitis
Acronym: PAROPAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PO15100
Record Dates: First submitted 2016-05-27; First posted 2016-06-08 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2017-03

CONDITIONS: Periodontal Disease : Chronic Periodontitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diseased (Other): Patients suffering of moderate to severe chronic periodontitis
  Interventions: Other: periodontal smears
- Healthy (Other): Healthy Patients not suffering of any periodontal disease a
  Interventions: Other: periodontal smears

INTERVENTIONS:
Other: periodontal smears

SUMMARY:
Periodontal diseases are complex chronic pathologies presenting a high prevalence worldwide. Etiopathological process involved in initiation and progression of these multifactorial diseases are not well understood, explaining the huge clinical forms variability and the complexity of the currently used classification of periodontal diseases. Recently, the implication of antimicrobial peptides (AMPs) have been suggested as potential track of explanation for periodontal diseases pathogeny. The here presented study explore the level of expression of genes coding those peptides by studying periodontal smears obtained from healthy and periodontitis patients.

DETAILED DESCRIPTION:
This study explore the level of expression of genes coding those peptides by studying Messenger RNA (mRNA) purified from periodontal smears obtained from healthy and periodontitis patients by "Masterpure©" protocol.After reverse transcription (RT-PCR), in-silico design of primers and specificity and efficiency calculation, Complementary DNA (cDNA) are quantified by a semi-quantitative method (delta-delta CT) vs a Housekeeping gene. Wilcoxon-Mann & Whitney tests and Chi² tests are performed to check the significativity of the results between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering of moderate to severe chronic periodontitis as described by the classification Armitage-1999, aged 35-65yo

Exclusion Criteria:

* Pregnant females, patients suffered from any other systemic diseases (cardiovascular, pulmonary, liver, cerebral, diseases or diabetes, cancer)
* patients that had received antibiotic treatment in the previous 3 months or who were taking long-term anti-inflammatory drugs; who had received a course of periodontal treatment or orthodontics treatment within the last 6 months; who were heavy smokers (>5 cig/day)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2016-03-23 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Antimicrobial peptides expression levels | Day 0
  Level of expression of antimicrobial peptides assessed by RT-PCR

SECONDARY OUTCOMES:
mRNA quantity | Day 0
  Quantity of mRNA purified on the smears

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France

REFERENCES:
- [Background] Jourdain ML, Pierrard L, Kanagaratnam L, Velard F, Sergheraert J, Lefevre B, Gangloff SC, Braux J. Antimicrobial peptide gene expression in periodontitis patients: A pilot study. J Clin Periodontol. 2018 May;45(5):524-537. doi: 10.1111/jcpe.12879. Epub 2018 Mar 23. PMID 29446150